## 07/17/2020

The Effect in Renal Function and Vascular Decongestion in Type 1 Cardiorenal Syndrome Treated with Two Strategies of Diuretics, a Randomized Clinical Trial

NCT04393493

## Statistical analysis

Based on the Shapiro-Wilk test, continuous variables are reported as the means (standard deviation [SD]) if they were normally distributed, or medians (interquartile range [IQR]) if they were not normally distributed. These variables were compared between groups with Mann-Whitney or t-tests as appropriate. Categorical variables are expressed as proportions and were compared by  $x^2$  tests or Fisher's exact test. For all tests, p values were two-sided, and a value <0.05 was considered statistically significant. MedCalc Statistical Software (Ostend, Belgium. Ver 19.1.3) was used for statistical analysis and graphics.